CLINICAL TRIAL: NCT06013696
Title: The Effect of Household Bleach on Urine Color Among Pediatric Ulcerative Colitis Patients Treated With 5-aminosalicylic Acid
Brief Title: Bleach and Urine Color in UC Patients Using 5ASA
Acronym: Asableach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, eyal zifman, Head of pediatric gastroenterology service, Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MMC-22-198
Record Dates: First submitted 2023-08-07; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Ulcerative Colitis
Keywords: Hematuria; Urine; 5-Aminosalycilic acid
MeSH Terms: conditions — Colitis, Ulcerative; Hematuria

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric UC subjects treated with 5ASA compunds (Active Comparator): Each subject will provide a fresh urine sample in an empty sterile plastic cup. Urinalysis will be performed to check for macro- or micro-hematuria or signs of infection. We will take 10mL of the urine sample and add 1mL of transparent (colorless) household bleach (≤5% sodium hypochlorite). The color of the urine before and 5 minutes after adding the bleach will be recorded.
  Interventions: Other: Adding household bleach to urine sample
- Pediatric UC subjects not treated with 5ASA compunds (any other treatments is allowed) (Placebo Comparator): Each subject will provide a fresh urine sample in an empty sterile plastic cup. Urinalysis will be performed to check for macro- or micro-hematuria or signs of infection. We will take 10mL of the urine sample and add 1mL of transparent (colorless) household bleach (≤5% sodium hypochlorite). The color of the urine before and 5 minutes after adding the bleach will be recorded.
  Interventions: Other: Adding household bleach to urine sample

INTERVENTIONS:
Other: Adding household bleach to urine sample — Adding household bleach to urine sample

SUMMARY:
The aim of this study is to evaluate the effect on urine color by adding household bleach to fresh urine sample among pediatric UC subjects treated with 5ASA

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect on urine color by adding household bleach to fresh urine sample among pediatric UC subjects treated with 5ASA.

ELIGIBILITY:
Inclusion Criteria:

1. UC patients in remission

Exclusion Criteria:

1. Acute UC exacerbation defined as Pediatric ulcerative colitis activity index (PUCAI) ≥10
2. Any acute or chronic renal disease, either present or past
3. Chronic hypertension, either present or past
4. Regularly receiving other medication that may cause nephrotoxicity - Non-steroidal anti-inflammatory drugs, acetaminophen, anti-epileptics, and antibiotics.
5. Pregnancy

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-16 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change is urine color | 5 minutes
  Following the addition of 1mL of 5% household bleach to a 10mL of each subject's urine, we will visually look for color change to red or orange within 5 minutes. Urine changing color to red or orange will be marked as a positive response to the bleach, which would fulfill the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Zifman, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No
According to instructions from our IRB the study's IPD is not to be shared. Specific requests may be sent after the study's completion and will be considered by the IRB .